CLINICAL TRIAL: NCT01085461
Title: Assessment of Suicidality in Epilepsy - Rating Tools
Acronym: ASERT
Status: Completed | Type: Observational
Sponsor: The Epilepsy Study Consortium (Other)
Collaborators: Eisai Inc. (Industry); GlaxoSmithKline (Industry); Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry); H. Lundbeck A/S (Industry); Pfizer (Industry); Supernus Pharmaceuticals, Inc. (Industry); UCB Pharma (Industry); Upsher-Smith Laboratories (Industry)
Responsible Party: Jacqueline French, MD, The Epilepsy Study Consortium
Other Study IDs: TESC-002
Record Dates: First submitted 2010-03-10; First posted 2010-03-11 (Estimated); Last update posted 2012-03-05 (Estimated); Status verified 2012-03

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
This will be a cross-sectional study enrolling 200 outpatients/inpatients with treatment resistant partial epilepsy for at least two years, receiving 1-3 AEDS.

The study will consist of one or two visits, each lasting 1-2 hours. All subjects will complete Visit 1. Twenty five percent of the subjects will return for Visit 2. The study will assess the prevalence of depression and suicidal thoughts and the feasibility of using the proposed psychiatric rating scales in future epilepsy clinical trials. This study will also provide an estimate of the proportion of patients with epilepsy (PWE) who may be ineligible for future trials.

DETAILED DESCRIPTION:
In light of the recent issues regarding antiepileptic drugs and suicidality, The Epilepsy Study Consortium is proposing a pilot study. Several scales to assess suicidality and screen for depression and anxiety disorders will be administered to a group of epilepsy patients with characteristics similar to patients who are usually enrolled in epilepsy clinical trials. The study will assess the prevalence of depression, suicidal thoughts, and behavior and the feasibility of using the proposed psychiatric rating scales in future epilepsy clinical trials. This study will also provide an estimate of the proportion of patients with epilepsy who may be ineligible for future trials because they have had active suicidal thoughts in the last 6 months, suicidal behavior in the last 2 years or a current major depressive episode.

ELIGIBILITY:
Inclusion criteria:

* Partial epilepsy for at least two years, confirmed with EEG studies
* Aged 18 to 70 years-old
* Proficient in English
* Having a minimum of a 4th grade reading level
* Having been on stable doses and type of AEDs for the previous two months
* Have at least 1 observable partial seizure (simple partial with motor component, complex partial or secondarily generalized tonic clonic seizure) per month for the past 6 months
* Is currently receiving 1-3 AEDs
* Has failed at least 2 AEDs (including current therapy)

Exclusion criteria:

* Non-epileptic seizures with or without comorbid epileptic seizures
* Subjects who currently carry a diagnosis of a major psychotic disorder
* Subjects who are currently taking an investigational medication
* Subjects with a known history of alcoholism, drug abuse, or drug addiction within the past 2 years

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with partial epilepsy for at least two years, who are treatment resistant, experience at least 1 seizure/month, and are receiving 1-3 AEDs/month will be selected.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2010-01; Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline French, M.D., Principal Investigator — NYU Langone Medical Center; Andres Kanner, M.D., Principal Investigator — Rush University Medical Center; Dale Hesdorffer, PhD, MPH, Principal Investigator — Columbia University; Kelly Posner, PhD, Principal Investigator — Columbia University
Locations (6):
- United States (6):
  - The International Center for Epilepsy (ICE) at the University of Miami, Miami, Florida
  - Rush Epilepsy Center, Chicago, Illinois
  - Johns Hopkins Hospital, Adult Epilepsy Center, Baltimore, Maryland
  - NYU Comprehensive Epilepsy Center, New York, New York
  - The Penn Epilepsy Center, Philadelphia, Pennsylvania
  - Jefferson Comprehensive Epilepsy Center, Philadelphia, Pennsylvania

REFERENCES:
- See also: The Epilepsy Study Consortium — http://www.epilepsyconsortium.org